CLINICAL TRIAL: NCT02553798
Title: An Open-label Study Assessing Long-term Safety of Glycopyrronium in Subjects With Primary Axillary Hyperhidrosis
Brief Title: Long-term Safety Study of Glycopyrronium in Subjects With Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRM04-HH06
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glycopyrronium (Experimental): Glycopyrronium Topical Wipes
  Interventions: Drug: Glycopyrronium Topical Wipes

INTERVENTIONS:
Drug: Glycopyrronium Topical Wipes — Glycopyrronium Topical Wipes
  Other Names: DRM04

SUMMARY:
This is an open-label, long-term safety study of glycopyrronium topical wipes, enrolling up to 660 subjects with primary axillary hyperhidrosis who participated in either the DRM04-HH04 or DRM04-HH05 studies.

DETAILED DESCRIPTION:
Safety will be assessed through adverse events, blood and urine laboratory tests, physical examination, pulse and blood pressure. Local skin reactions will be assessed including burning/stinging, pruritus, edema, erythema, dryness and scaling.

ELIGIBILITY:
Inclusion Criteria:

* Completed Day 28 of either the DRM04-HH04 or DRM04-HH05 study with at least 80% treatment compliance
* Male or females

Exclusion Criteria:

* Subject has a clinically significant abnormality on physical exam, vital signs or ECG at the Week 4 visit of DRM04-HH04 or DRM04-HH05 study that would make further treatment with glycopyrronium contraindicated
* Male with a history of urinary retention requiring catheterization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy
* Any other condition which, in the judgement of the Investigator, would put the subject at unacceptable risk for participation in the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Deans, MT, Study Director — Dermira, Inc.
Locations (48):
- United States (40):
  - Coastal Medical Research Group LLC, Mobile, Alabama
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Colorado Medical Research Center, Inc, Denver, Colorado
  - Skin Care Research, Inc., Boca Raton, Florida
  - Study Protocol, Inc, Boynton Beach, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Tory Sullivan, MD, North Miami Beach, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Prairie Health and Wellness, Wichita, Kansas
  - Lawrence J. Green M.D., LLC, Rockville, Maryland
  - Zel Skin & Laser Specialist, Edina, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - St. Louis University Dermatology, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Schweiger Dermatology Group, New York, New York
  - Skin Search of Rochester, Inc, Rochester, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology and Laser Center of Charleston, PA, Charleston, Pennsylvania
  - Rivergate Dermatology Research Center, PLLC, Goodlettsville, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - DermResearch, Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - The University of Texas Dermatology Clinical Research Center, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - ACRC Trials, Plano, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Jordan Valley Dermatology Center, LLC, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Germany (8):
  - Klinik für Dermatologie, Venerologie und Allergologie Allergie-Centrum-Charité, Berlin
  - Pro DERMA im Hautzentrum Dulmen, Dülmen
  - Medical Practice and Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Hautarztpraxis, Glückstadt
  - Tagesklinik DermaKiel, Kiel
  - Dermatolosche Gemeinschaftspraxis, Mahlow
  - Gemeinschaftspraxis Weber & Cranic, Schweinfurt

REFERENCES:
- [Derived] Glaser DA, Hebert AA, Nast A, Werschler WP, Green L, Mamelok RD, Quiring J, Drew J, Pariser DM. A 44-Week Open-Label Study Evaluating Safety and Efficacy of Topical Glycopyrronium Tosylate in Patients with Primary Axillary Hyperhidrosis. Am J Clin Dermatol. 2019 Aug;20(4):593-604. doi: 10.1007/s40257-019-00446-6. PMID 31111409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glycopyrronium
Started | 564
Completed | 226
Not Completed | 338

BASELINE CHARACTERISTICS:
Arm/Group | Glycopyrronium
Number analyzed (Participants) | 564
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 499
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309
  Male | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97
  Not Hispanic or Latino | 467
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 64
  White | 470
  More than one race | 24
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety Assessed Through Adverse Events and Local Skin Reactions
Description: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Time Frame: Day 1 - Week 44
Population: Participant
Measure: Number; unit: Adverse Events and Local Skin Reactions
Arm/Group | Glycopyrronium
Number analyzed (Participants) | 550
Adverse Events and Local Skin Reactions
  Mild AEs | 148
  Moderate AEs | 153
  Severe AEs | 28
  Mild LSRs | 120
  Moderate LSRs | 44
  Severe LSRs | 15

2. Other Pre Specified Outcome: Mean Absolute Change From Baseline in Gravimetrically-measured Sweat Production at Week 4
Description: Subjects are acclimated to the environment for 30 minutes. Dry gauze is weighed. The dry gauze is then applied to the subject's axilla with the arm down by the subject's side or on their lap during the 5-minute period of sweat production. The gauze with the sweat is then weighed. The difference between the Weight of the gauze with sweat and the dry gauze is the gravimetric sweat measurement in mg/5min.
Time Frame: Baseline (from DRM04-HH04 (NCT02530281) or DRM04-HH05 (NCT02530294) study) - Week 44/ET
Population: Participant
Measure: Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Glycopyrronium
Number analyzed (Participants) | 430
mg/5 min | -95.68 (140.806)

3. Other Pre Specified Outcome: Grade Improvement in Hyperhidrosis Disease Severity Scale (HDSS)
Description: Hyperhidrosis Disease Severity Scale (HDSS) is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.
Time Frame: Baseline (from DRM04-HH04 (NCT02530281) or DRM04-HH05 (NCT02530294) study) - Week 44/ET
Population: Participant
Measure: Number; unit: participants
Arm/Group | Glycopyrronium
Number analyzed (Participants) | 437
participants
  3 - point improvement | 72
  2 - point improvement | 204
  1 - point improvement | 135
  no improvement | 26

4. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 44/ET
Description: The Dermatology Life Quality Index DLQI is a ten question questionnaire, used to measure the impact of skin disease on the quality of life of an affected person. The scoring of each question is as follows: Very much (3), A lot (2), A little (1), Not at all (0), Not relevant (0). Is calculated by summing the score of each question resulting in a max of 30 and a min of 0. Higher the score the more Quality of life is impaired.
Time Frame: Baseline (from DRM04-HH04 (NCT02530281) or DRM04-HH05 (NCT02530294) study) - Week 44/ET
Population: Participant
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Glycopyrronium
Number analyzed (Participants) | 406
scores on a scale | -8.7 (6.24)

ADVERSE EVENTS:
Time Frame: up to 45 weeks
Description: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Glycopyrronium
All-Cause Mortality (participants affected / at risk) | 0/550
Serious Adverse Events (participants affected / at risk) | 7/550
Other Adverse Events (participants affected / at risk) | 178/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium (N=550)
Diverticulitis (Infections and infestations) | 1
Infectious colitis (Infections and infestations) | 1
Affective disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Mydriasis (Eye disorders) | 1
Chest pain (General disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium (N=550)
Dry Mouth (Gastrointestinal disorders) | 93
Nasopharyngitis (Infections and infestations) | 32
Application Site Pain (General disorders) | 35
Vision blurred (Eye disorders) | 37
Mydriasis (Eye disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes